CLINICAL TRIAL: NCT06692049
Title: Gonadal Tissue Cryopreservation for Fertility Preservation in Children with a Disorder of Sex Development
Acronym: DSD
Status: Recruiting | Type: Observational
Sponsor: Erin Rowell (Other)
Collaborators: Ann & Robert H Lurie Children's Hospital of Chicago (Other)
Responsible Party: Sponsor-Investigator, Erin Rowell, Director, Fertility & Hormone Preservation & Restoration, Ann & Robert H Lurie Children's Hospital of Chicago
Organization: Ann & Robert H Lurie Children's Hospital of Chicago (Other)
Other Study IDs: 2017-1164
Record Dates: First submitted 2020-08-28; First posted 2024-11-18 (Actual); Last update posted 2024-11-18 (Actual); Status verified 2024-11

CONDITIONS: DSD, 46,XY; DSD, Ovotesticular; DSD, Sex Chromosome; Disorders of Sex Development; Disorder of Sex Development, 46,XY; Disorder of Sex Development, 46,Xy, Cbx2-Related
Keywords: DSD; GTC; Gonadectomy; Cryopreservation; Fertility Preservation
MeSH Terms: conditions — Disorder of Sex Development, 46,XY; Ovotesticular Disorders of Sex Development; Sex Chromosome Disorders of Sex Development; Disorders of Sex Development; 46, XY Sex Reversal 5 | interventions — Castration

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Biospecimen Retention: Samples With DNA — Tissue and blood specimens collected
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Disorders of Sex Development (DSD): The study seeks to find out if removing gonadal tissue in adolescents and children at risk for losing fertility potential (the ability to have children) and who are scheduled to receive a gonadectomy (removal of gonads) for clinical purposes may preserve, or keep, their ability to have children in the future. Additionally, donated research tissue would be used to study long-term ways to preserve and restore reproductive function of children diagnosed with DSD
  Interventions: Procedure: Gonadectomy

INTERVENTIONS:
Procedure: Gonadectomy — Gonadal tissue being removed for risk of malignancy may be cryopreserved for fertility preservation

SUMMARY:
The purpose of this study is to offer gonadal tissue freezing and storage to children who are diagnosed with a disorder of sex development (DSD), who are at increased risk of infertility and certain malignancies (cancer). This study involves the storage of gonadal tissue that is being removed for medical reasons (e.g. prevention of cancer development). It includes the processing and freezing of this gonadal tissue, hopefully for potential future use. The tissue will then be stored long-term until the child wishes to try to use the tissue.

DETAILED DESCRIPTION:
DSD are conditions in which there is incongruence in an individual's chromosomal, gonadal, or phenotypic sex (refers to sex as determined by an individual's internal or external genitalia and expression of secondary sex characteristics).Different DSD diagnoses have varying degrees of risk for future malignancy. The treating doctor has or will discuss with the participant the risk of developing cancer due to the child's specific diagnosis, and help decide whether this option is in the best interest of the child, and if there are other options to consider (e.g. leaving gonadal tissue in place and monitoring for development of malignancy). If the participant and family have decided to move forward with removal of gonadal tissue for this clinical reason, they will be asked if they would like to have the child participate in this study.

This study seeks to find out if removing gonadal tissue in adolescents and children at risk for losing fertility potential (the ability to have children) and who are scheduled to receive a gonadectomy (removal of gonads) for clinical purposes may preserve, or keep, their ability to have children in the future. Additionally, a primary objective of this study is to use donated research tissue to study long-term ways to preserve and restore reproductive function for children diagnosed with a DSD. Gonadal tissue cryopreservation in patients diagnosed with a DSD is still considered experimental. There have been no reported live births or pregnancies in this population following gonadal tissue cryopreservation at this time.

ELIGIBILITY:
Inclusion Criteria:

* Individual < 30 years of age
* Children diagnosed with a disorder of sex development who have any risk for malignancy in their gonadal tissue or will have their gonads removed for another clinical indication

Exclusion Criteria:

* Pregnant children
* Patients likely to retain inherent fertility and reproductive function
* Children deemed high risk for perioperative complications
* Patients 12-18 unable to provide assent (i.e. significant psychiatric problems/cognitive delay)
* Patients 18 and older unable to provide consent (i.e. significant psychiatric problems/cognitive delay)

Max Age: 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Children diagnosed with a disorder of sex development who have any risk for malignancy in their gonadal tissue or will have their gonads removed for another clinical indication
Sampling Method: Non-Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2018-04-04 (Actual); Primary Completion 2030-12-31 (Estimated); Study Completion 2035-12-31 (Estimated)

PRIMARY OUTCOMES:
Gonadal Tissue Cryopreservation for Fertility Preservation in Children with Disorders of Sex Development | 3 months
  The primary outcome is histologic evaluation of the gonads for the presence of germ cells which will be cryopreserved for potential future fertility.

SECONDARY OUTCOMES:
Gonadal Tissue Cryopreservation for Fertility Preservation in Children with Disorders of | yearly, up to 20 years
  Secondary outcomes include long term follow up of study participants for development of secondary sex characteristics, puberty progression, and ability for the participant to have their own children as adults if desired.

CONTACTS AND LOCATIONS:
Overall Officials: Erin Rowell, MD, Principal Investigator — Ann & Robert H Lurie Children's Hospital of Chicago
Locations (1):
- Ann & Robert H. Lurie Children's Hospital of Chicago, Chicago, Illinois, United States